CLINICAL TRIAL: NCT02685891
Title: Exploring Diurnal Changes in Markers of Cortical Plasticity Using Multimodal Imaging in Healthy Children, Adolescents and Adults
Brief Title: Brain Maturation and Sleep
Acronym: BMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PB_2016-00254
Record Dates: First submitted 2016-02-04; First posted 2016-02-19 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- playing tones (Active Comparator): During slow-wave sleep short tones (50ms, 50dB) will be played
  Interventions: Other: Playing tones during deep sleep
- Playing no tones (Sham Comparator): During slow-wave sleep no tones will be played
  Interventions: Other: sham condition

INTERVENTIONS:
Other: Playing tones during deep sleep — Playing tones time locked to slow waves (Duration:50ms, volume: 50dB)
  Arms: playing tones
Other: sham condition — in the sham condition, no tones will be played
  Arms: Playing no tones

SUMMARY:
In this study, the investigator evaluates whether there are age-specific diurnal changes in markers of cortical plasticity in children, adolescents and adults. The question will be investigated by the quantification of brain metabolites and structural brain volumes using magnet resonance imaging (MRI) and electrophysiological markers using sleep encephalography (sleep EEG). In a second step, it will be tested how these markers of cortical plasticity change depending on a modulation of sleep by applying tones during deep sleep.

DETAILED DESCRIPTION:
Given that children and adolescents undergo entirely different maturational processes (children show an increase, adolescents a decrease in synapse density) larger diurnal changes in children are expected compared to adolescents concerning brain metabolites and structural markers. These cortical changes in synapse density are thought to be reflected in electrophysiological markers in the sleep EEG (children show a higher slow wave activity, adolescents a reduced slow wave activity). With the modulation of the deep (slow wave) sleep by playing short, low volume tones, the investigators want to test if there is a causal relationship between slow wave sleep and markers of cortical plasticity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 8 to 30 years of age,
* good general health Status
* right-handedness,
* Written informed consent after participants' information

Exclusion Criteria:

* sleep disorders (insomnia, sleep disordered breathing, restless legs syndrome)
* sleep complaints in general
* irregular sleep-wake rhythm
* daytime sleep
* travelling across a time zone within the last month
* diseases or lesions of the central nervous system
* psychiatric diseases
* learning disability
* skin allergy or very sensitive skin
* acute pediatric disease
* pregnancy
* drug and medication use and abuse
* nicotine use
* high caffeine consumption (>2 servings/day (>160 mg caffeine); including coffee, tea, white and dark chocolate, coca cola, energy drink)
* Alcohol consumption in children and adolescents under 16 years
* high alcohol consumption in adults (> 1 standard serving/day (>14 mg Alcohol))
* high alcohol consumption in adolescents aged 16 years and above (> 3-4 Standard servings per week)

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-06; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diurnal changes in brain metabolites | 3 years
  concentration of brain metabolites measured by MR spectroscopy change from evening to morning

SECONDARY OUTCOMES:
electrophysiological markers change in dependance of the diurnal variation of brain metabolites | 3 years
  electrophysiological markers (sleep EEG) change in dependance of the diurnal variation of brain metabolites
structural markers change in dependance of the diurnal variation of brain metabolites | 3 years
  structural markers (MR volumes) change in dependance of the diurnal variation of brain metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland